CLINICAL TRIAL: NCT01904032
Title: Vitamin D Supplement to Women With Type 2 Diabetes
Brief Title: Sunshine 2 Study for Women With Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sue, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 204197; 1R01NR013906-01A1 (NIH)
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-03

CONDITIONS: Diabetes; Depression; Quality of Life
Keywords: Vitamin D; Diabetes; Self-Management; Depression; Women
MeSH Terms: conditions — Diabetes Mellitus; Depression | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either 50,000 international units of weekly vitamin D3 or to 5,000 international units of weekly vitamin D3 using a 1:1 allocation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 (Experimental): 50,000 international units (IUs) weekly Vitamin D3
  Interventions: Drug: Vitamin D3
- Vitamin D3 comparator (Active Comparator): 5,000 international units (IUs) of a weekly Vitamin D3 comparator
  Interventions: Drug: Vitamin D3 comparator

INTERVENTIONS:
Drug: Vitamin D3 — 50,000 international units (IUs) weekly Vitamin D3
  Other Names: Cholecalciferol
  Arms: Vitamin D3
Drug: Vitamin D3 comparator — 5,000 international units (IUs) of a weekly Vitamin D3 comparator
  Other Names: Cholecalciferol
  Arms: Vitamin D3 comparator

SUMMARY:
This is a randomized clinical trial (RCT) to determine the effectiveness of vitamin D3 supplementation on depressive symptoms, self-management, and blood pressure in approximately 180 adult women with type 2 diabetes who have significant depressive symptoms. Consenting adult women who are eligible to participate will be randomly assigned to either a weekly dose of 50,000 international units of vitamin D3 supplementation or a matching weekly active comparator of 5,000 international units of vitamin D3 for six months. Participants will complete approximately four in-person study visits and several telephone visits throughout the six month trial period, where the researchers will assess depressive symptoms, diabetes self-management, and systolic blood pressure.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the effect of vitamin D supplementation on depressive symptoms, self-management, and systolic blood pressure compared to placebo. The hypothesis is that women receiving vitamin D supplementation will report fewer depressive symptoms, increased diabetes self- management mediated by depression improvement, and will have a lower systolic blood pressure compared to those taking placebo at three and six months follow-up.

The secondary aim is to explore the mechanistic effect of vitamin D supplementation on inflammatory biomarkers and their association with depression. Here, the hypothesis is that women receiving vitamin D supplementation will have a decrease in inflammatory biomarkers which will be associated with fewer depressive symptoms compared to those taking placebo at three and six months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women age 21 and older
* Objective evidence of depressive symptoms at the screening and baseline visits
* Diagnosis of type 2 diabetes currently being treated by a healthcare provider
* Blood vitamin D level less than 32 nanograms-per-deciliter (32 ng/dl)

Exclusion Criteria:

* Current alcohol or substance use disorder
* Any unstable or severe psychiatric disease including diagnoses of schizophrenia, bipolar affective disorder, dementia, delirium, or other psychotic disorder
* Severe complications of diabetes, such as blindness and/or amputation
* Any malabsorption disorder, such as Crohn's disease and/or celiac sprue
* Elevated serum calcium level deemed significant by the Principal Investigator
* Use of 1,000 or more international units daily vitamin D 60 days before enrollment and unwillingness to discontinue vitamin D supplementation 30 days before enrollment.
* Use of St. John's Wort and unwillingness to discontinue St. John's Wort three weeks prior to enrollment.
* Participants who are pregnant, nursing, or planning to become pregnant during the study.
* Baseline systolic blood pressure (SBP) greater than 160 millimeters of mercury (mmHG) or diastolic blood pressure (DBP) greater than 100 mmHG.
* Other serious medical conditions (e.g., cancer, multiple sclerosis, etc.) deemed clinically significant by the Principal Investigator

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Penckofer, Ph.D., R.N., Principal Investigator — Loyola University Chicago Health Sciences Division
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from November 2013 through November 2017 (48 months)
Pre-assignment Details: Two-hundred sixty-five participants consented to participate in the study. Among these individuals, 136 (51.3%) were not randomized for failing to meet study inclusion criteria (134/136 or 98.5%) or because they withdrew consent prior to randomization (2/136 or 1.5%).
Groups:
- Low Dose: 5,000 international units (IUs) of a weekly Vitamin D3 comparator
- High Dose: 50,000 international units (IUs) weekly Vitamin D3
Period: Overall Study
Arm/Group | Low Dose | High Dose
Started | 64 | 65
Completed | 57 | 62
Not Completed | 7 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all patients randomized to high dose or lose dose therapy
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.14 (9.40) | 50.02 (12.65) | 50.58 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 129
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 23
  Not Hispanic or Latino | 53 | 53 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 34 | 29 | 63
  Race: Black | 28 | 34 | 62
  Race: Asian or Pacific Islander | 1 | 1 | 2
  Race: Arabic | 0 | 1 | 1
  Race: Not reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 64 | 65 | 129
Use of anti-depressants [Count of Participants; unit: Participants]
  No | 53 | 52 | 105
  Yes | 11 | 12 | 23
  Not reported | 0 | 1 | 1
Highest level of education [Count of Participants; unit: Participants]
  8th grade or less | 0 | 1 | 1
  Some high school | 5 | 2 | 7
  High school graduate or GED | 10 | 8 | 18
  Some college or technical school | 24 | 26 | 50
  College graduate (bachelor's degree) | 16 | 17 | 33
  Graduate degree | 9 | 11 | 20
Annual Household Income [Count of Participants; unit: Participants]
  Less than $5,000 | 5 | 7 | 12
  $5,000 to $9,999 | 4 | 4 | 8
  $10,000 to $14,999 | 9 | 4 | 13
  $15,000 to $19,999 | 1 | 5 | 6
  $20,000 to $29,999 | 5 | 9 | 14
  $30,000 to $39,999 | 8 | 5 | 13
  $40,000 to $49,999 | 5 | 9 | 14
  $50,000 to $59,999 | 6 | 6 | 12
  $60,000 to $69,999 | 4 | 4 | 8
  $70,000 or more | 17 | 12 | 29
CES-D [Mean (Standard Deviation); unit: units on a scale] — The Center for Epidemiologic Studies Depression (CES-D) score is a self-report questionnaire assessing frequency and severity of depression symptoms. Scores may range from 0 to 60, where higher scores indicate worse mood.
  units on a scale | 28.41 (8.39) | 28.72 (8.50) | 28.57 (8.41)
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ) is a self-administered depression screening inventory. Scores range from 0 to 27 with higher scores indicating worse mood
  units on a scale | 11.91 (4.20) | 11.74 (4.29) | 11.82 (4.23)
Vitamin D3 Level [Mean (Standard Deviation); unit: ng/mL] | 18.61 (6.66) | 20.63 (6.60) | 19.63 (6.68)
Parathyroid Hormone [Median (Inter-Quartile Range); unit: ng/L] | 49 [36 to 69] | 49 [38 to 59] | 49 [36 to 64]
Calcium [Median (Inter-Quartile Range); unit: mg/dL] | 9.4 [9.2 to 9.7] | 9.4 [9.2 to 9.6] | 9.4 [9.2 to 9.6]
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.74 (0.14) | 0.75 (0.15) | 0.75 (0.14)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 128.41 (16.40) | 127.43 (14.96) | 127.91 (15.63)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 71.97 (10.64) | 70.94 (8.75) | 71.45 (9.71)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 39.10 (8.28) | 37.65 (7.71) | 38.37 (8.00)
HBA1C [Mean (Standard Deviation); unit: percentage of hemoglobin] | 7.86 (1.97) | 7.68 (1.69) | 7.77 (1.83)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 170.47 (68.63) | 152.52 (48.76) | 161.43 (59.90)

OUTCOME MEASURES:

1. Primary Outcome: Change in Center for Epidemiologic Studies Depression (CES-D) Score From Baseline (Month 0) to Month 6 for the High Dose Cohort Versus Low Dose Cohort
Description: The Center for Epidemiologic Studies Depression (CES-D) is a self-report questionnaire assessing frequency and severity of depression symptoms. Raw scores range from 0 to 60, where higher scores indicate worse mood. For each participant, her baseline CES-D score is subtracted from her month 6 CES-D score to create a CES-D change score.
Time Frame: Baseline and 6 months
Population: The analysis population includes all women randomized to low dose or high dose therapy and completed the month 6 CES-D assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 57 | 62
units on a scale | -13.2982 (10.2312) | -12.5000 (12.0065)
Statistical Analysis 1: Comparison: Low Dose vs High Dose; The null hypothesis is that there is no difference in the CES-D change score between women who received high dose Vitamin D therapy versus low dose Vitamin D therapy; Test type: Superiority; p = .6982, t-test, 2 sided; Mean Difference (Final Values) = 0.7982, 95% CI 2-sided [-3.2691 to 4.8656], Standard Error of Mean 2.0537

2. Secondary Outcome: Change in Problem Areas in Diabetes (PAIDS) Score From Baseline (Month 0) to Month 6 for the High Dose Cohort Versus Low Dose Cohort
Description: The Problem Areas in Diabetes (PAIDS) score is a self-report questionnaire that assesses diabetes burden and treatment. Scores range from 0 to 100, where higher scores indicate greater distress. For each participant, her baseline PAID score is subtracted from her month 6 PAID score to create a PAID change score.
Time Frame: Baseline and 6 months
Population: The analysis population includes all women randomized to low dose or high dose therapy and completed the month 6 PAID assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 57 | 62
score on a scale | -13.2237 (17.6238) | -13.2661 (21.8782)
Statistical Analysis 1: Comparison: Low Dose vs High Dose; The null hypothesis is that there is no difference in the PAID change score between women who received high dose Vitamin D therapy versus low dose Vitamin D therapy; Test type: Superiority; p = .9908, t-test, 2 sided; Mean Difference (Final Values) = -0.0424, 95% CI 2-sided [-7.2946 to 7.2097], Standard Error of Mean 3.6619

3. Secondary Outcome: Change in Systolic Blood Pressure From Baseline (Month 0) to Month 6 for the High Dose Cohort Versus Low Dose Cohort
Description: Systolic blood pressure is measured in millimeters of mercury (mmHg). For each participant, her baseline systolic blood pressure is subtracted from her month 6 systolic blood pressure to create a systolic blood pressure change score.
Time Frame: Baseline and 6 months
Population: The analysis population includes all women randomized to low dose or high dose therapy and completed the in-person month 6 study visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 57 | 62
mmHg | -2.1579 (17.6491) | -1.6613 (16.6821)
Statistical Analysis 1: Comparison: Low Dose vs High Dose; The null hypothesis is that there is no difference in the change in systolic blood pressure between women who received high dose Vitamin D therapy versus low dose Vitamin D therapy; Test type: Superiority; p = .8749, t-test, 2 sided; Mean Difference (Final Values) = 0.4966, 95% CI 2-sided [-5.7366 to 6.7298], Standard Error of Mean 3.1474

4. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline (Month 0) to Month 6 for the High Dose Cohort Versus Low Dose Cohort
Description: Diastolic blood pressure is measured in millimeters of mercury (mmHg). For each participant, her baseline diastolic blood pressure is subtracted from her month 6 diastolic blood pressure to create a diastolic blood pressure change score.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 57 | 62
mmHg | -0.7544 (10.6692) | 0.7581 (9.6609)
Statistical Analysis 1: Comparison: Low Dose vs High Dose; The null hypothesis is that there is no difference in the change in diastolic blood pressure between women who received high dose Vitamin D therapy versus low dose Vitamin D therapy; Test type: Superiority; p = .4187, t-test, 2 sided; Mean Difference (Final Values) = 1.5125, 95% CI 2-sided [-2.1784 to 5.2033], Standard Error of Mean 1.8636

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for seven months
Arm/Group | Low Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/65
Serious Adverse Events (participants affected / at risk) | 5/64 | 7/65
Other Adverse Events (participants affected / at risk) | 55/64 | 60/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=64) | High Dose (N=65)
Right sided weakness (Nervous system disorders) | 0 (0) | 1 (1) — Right sided weakness resulting in an inpatient hospitalization
Stroke (Nervous system disorders) | 0 (0) | 1 (1) — Stroke resulting in an inpatient hospitalization
Acoustic neuroma (Nervous system disorders) | 0 (0) | 1 (1)
Severe abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) — Severe abdominal pain resulting in inpatient hospitalization
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Unplanned pregnancy considered an important medical event
Left tibia fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Left tibia fracture resulting in an inpatient hospitalization
Laparoscopic cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — Unplanned laparoscopic cholecystectomy resulting in an inpatient hospitalization
Hiatal Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hiatal hernia resulting in an inpatient hospitalization
Cancer Diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Right total knee replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unplanned right total knee replacement resulting in an inpatient hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=64) | High Dose (N=65)
Infection (Infections and infestations) | 16 (25) | 12 (17)
Joint Pain (Musculoskeletal and connective tissue disorders) | 17 (24) | 11 (14)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (8)
Generalized Pain (General disorders) | 1 (1) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 7 (8) | 7 (10)
Upper Respiratory Symptoms (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 7 (7)
Dizziness (General disorders) | 7 (9) | 3 (7)
Abnormal Kidney Function (Renal and urinary disorders) | 4 (8) | 3 (9)
Elevated Glucose (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 7 (7)
Nausea (General disorders) | 4 (5) | 11 (17)
Influenza (Infections and infestations) | 0 (0) | 5 (5)
Headache (General disorders) | 7 (7) | 7 (7)
Routine Surgery (Surgical and medical procedures) | 7 (9) | 3 (3)
Worsening Mood (Psychiatric disorders) | 17 (17) | 19 (19)
Worsening Diabetes (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Muscle Pain (General disorders) | 3 (4) | 4 (4)
Numbness (Nervous system disorders) | 4 (4) | 6 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Lower Extremity Cramps (General disorders) | 4 (4) | 2 (2)
Menstrual Symptoms (Reproductive system and breast disorders) | 0 (0) | 8 (8)
Fatigue (General disorders) | 5 (6) | 8 (8)
Generalized Soreness (General disorders) | 3 (4) | 4 (4)
Swelling (General disorders) | 1 (1) | 5 (5)
Fall (General disorders) | 11 (17) | 6 (6)
Hypertension (General disorders) | 6 (7) | 6 (8)

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT01904032/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT01904032/ICF_001.pdf